CLINICAL TRIAL: NCT03087695
Title: Effect of the Plasma EBV DNA Concentration Change During Chemoradiotherapy on Tumor Control and Patient Survival in Advanced Nasopharyngeal Carcinoma
Brief Title: Effect of the Plasma EBV DNA Change During Chemoradiotherapy in Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CF17002B
Record Dates: First submitted 2017-03-06; First posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; EBV DNA; Chemoradiotherapy
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The patients will be collected blood sample once per week during chemoradiotherapy period. Plasma will be extracted from these blood sample. Plasma EBV DNA concentrations will be measured by a real-time quantitative polymerase chain reaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Plasma EBV DNA — Parameters analyzed will include (1) the change pattern of plasma EBV DNA concentrations, (2) various half-life values (t1/2) of plasma EBV DNA clearance rate calculated over different time periods.

SUMMARY:
Epstein-Barr virus (EBV) has been proven to process a strong association in patient of nasopharyngeal carcinoma (NPC). Monitoring plasma EBV DNA in NPC patients can provide reliable informations in early detecting tumor recurrence or risk grouping.

DETAILED DESCRIPTION:
EBV DNA has strongly association in NPC patient' disease status. It can provide informations of disease relapse or risks classification. In this study, we will investigate the impact of plasma EBV DNA concentration change during chemoradiotherapy on initial tumor response and long-term survival in patients with advanced nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histological proven NPC.
2. 2010 American Joint Committee on Cancer (AJCC) stage II-IVB.
3. Age ≧ 20 years old.
4. Performance status of Eastern Cooperative Oncology Group (ECOG) ≦ 2.
5. Adequate liver, renal, and bone marrow functions 5.1 Serum total bilirubin level ≦ 2.5 mg/dl. 5.2 Serum creatinine ≦ 1.6 mg/dl or calculated creatinine clearance rate (CCr) ≧ 60 cc/min.

   5.3 White blood cell count (WBC) ≧ 3,000/micro-ml. 5.4 Platelet count ≧ 100,000/micro-ml.
6. Pre-treatment plasma EBV DNA > 0 copies/mL
7. Signed informed consent.

Exclusion Criteria:

1. Presence of distant metastasis.
2. Previous radiotherapy or chemotherapy.
3. History of a malignancy except those treated with curative intent for skin cancer (other than melanoma), in situ cervical cancer, ductal carcinoma in situ (DCIS) of the breast.
4. Severe cardiopulmonary diseases (unstable angina and/or congestive heart failure or peripheral vascular disease requiring hospitalization within the last 12 months; chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization) or clinically significant psychiatric disorders.
5. Female patients who are pregnant or lactating.

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Nasopharyngeal carcinoma patient received definite treatment in Taichung Veteran General Hospital
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-04-01 (Estimated); Primary Completion 2018-01-16 (Estimated); Study Completion 2019-01-16 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2 years
  Survival calculation

SECONDARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Survival calculation
Nasopharynx failure-free survival (NPFFS) | 2 years
  Survival calculation
Neck failure-free survival (NFFS) | 2 years
  Survival calculation
Distant metastasis failure-free survival (DMFFS) | 2 years
  Survival calculation
Tumor response | 2 years
  Tumor response evaluated by image
EBV DNA concentration | 2 years
  Plasma EBV DNA by real-time polymerase chain reaction (PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ching Lin, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (1):
- Taichung Veteran General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No
No plan to make individual participant data (IPD) available